"Evaluation of The Effect of Neck and Trunk Stabilization Exercises on Quality of Life and Communication in Children with Cerebral Palsy with Oral Motor Problem"

NCT04214080

23.03.2018

## STUDY PROTOCOL

## **Scientific Background:**

Trunk control of children with CP has been affected by spasticity, weakness in the trunk muscles, incoordination activation of trunk extensor and flexor muscles. Trunk stabilization exercises are an essential component of the mobility of distal part of body, including neck movements. Strengthening the deep neck flexor muscles and bridge exercise improves trunk control in children with CP. The positive effects of neck and trunk stabilization exercises on static and dynamic trunk balance, on upper limb and visuoperceptual function in CP have been mentioned in the literature.

## **Objectives:**

According to literature there was a relationship between vocal functions and posture, active trunk movements has an important role in sound production and lastly trunk stabilization, balance and activity level components are in relationship with each other. Thus in this study, it was aimed to investigate the effects of neck and trunk stabilization exercises on communication, activities of daily living and quality of life in children with CP with oral motor problem.

## Design:

The effects of structured neck and trunk stabilization exercises program giving together with feeding and oral-motor intervention strategies in children with Cerebral Palsy with oral motor problem: a randomized, single-blind, placebo controlled study. In this study, children were divided into study and control groups using a randomized numbers table. Structured oral motor rehabilitation and Neurodevelopmental therapy method-Bobath concept (NDT-B) approach was performed to all of the children who were in accordance with the inclusion criteria and approved by their families. In addition to the structured oral motor rehabilitation and NDT-B approach, *Study* group was received intensive structured neck and trunk stabilization exercises based on NDT-B principles.

| Sponsor: | Marmara University, Istanbul, Turkey |
|---|---|
| Measured Parameters: | -Gross motor functions, |
| | -Daily communication performance, |
| | -Speech production, |
| | -The capacity to do the activities in daily life, |
| | -The physical functions, psychosocial functions and school functionality independent of disease in children, |
| | -Evaluation of trunk in sitting position. |
| Study Center: | Marmara University Pendik Education And Research Hospital,<br>Istanbul, Turkey |

All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards. Ethical approval was obtained from the Marmara University Faculty of Medicine Clinical Research **Ethics Committee protocol code 09.2018.278.**